CLINICAL TRIAL: NCT03365362
Title: Achieving Smoking Cessation Milestones in Opioid Treatment Patients: a Randomized 2 x 2 Factorial Trial of Directly Observed and Long-term Varenicline
Brief Title: A Trial of Directly Observed and Long-term Varenicline
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Pfizer (Industry); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-6688; R01DA042813 (NIH)
Record Dates: First submitted 2017-11-28; First posted 2017-12-07 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Tobacco Use Disorder; Opioid-use Disorder
Keywords: directly observed therapy; varenicline; long-term pharmacotherapy
MeSH Terms: conditions — Tobacco Use Disorder; Opioid-Related Disorders; Directly Observed Therapy | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Long-Term Varenicline (Experimental): Participants will receive 24 weeks of varenicline at standard doses (0.5 mg/day for days 1 to 3, 0.5 mg twice daily for days 4 to 7, then 1 mg twice daily)
  Interventions: Drug: Long-Term Varenicline
- Short-Term Varenicline (Active Comparator): Participants will receive 12 weeks of varenicline at standard doses (0.5 mg/day for days 1 to 3, 0.5 mg twice daily for days 4 to 7, then 1 mg twice daily), followed by matching placebo twice daily through week 24.
  Interventions: Drug: Short-Term Varenicline
- Directly Observed Therapy (Experimental): Participants receiving directly observed therapy (DOT) will receive varenicline from opioid treatment program nurses at the same time as they receive methadone, as well as individually packaged take-home doses for self administration on evenings/weekends.
  Interventions: Behavioral: Directly Observed Therapy
- Self Administered Therapy (Active Comparator): Patients receiving varenicline self administered therapy (SAT) will self-administer all varenicline doses.
  Interventions: Behavioral: Self Administered Therapy

INTERVENTIONS:
Drug: Long-Term Varenicline — Varenicline tablet x 24 weeks
  Other Names: varenicline; chantix
  Arms: Long-Term Varenicline
Drug: Short-Term Varenicline — varenicline tablet for 12 weeks, followed by placebo tablet manufactured to mimic varenicline 1 mg tablet
  Other Names: varenicline; chantix; placebo
  Arms: Short-Term Varenicline
Behavioral: Directly Observed Therapy — Varenicline doses are administered by opioid treatment program nurses
  Arms: Directly Observed Therapy
Behavioral: Self Administered Therapy — Varenicline doses are self-administered
  Arms: Self Administered Therapy

SUMMARY:
This 2 x 2 factorial, randomized, double-blind, placebo-controlled trial will test two interventions: directly observed medication therapy, and long-term therapy with varenicline among smokers with opioid use disorder recruited from community-based, outpatient opioid treatment programs. The analytic strategy will evaluate the milestones in smoking cessation-achieving initial abstinence, preventing lapse and preventing relapse--necessary for long-term cessation, and evaluate theoretically-guided psychological and social factors and pharmacogenetic factors that influence these cessation processes.

DETAILED DESCRIPTION:
Tobacco use and tobacco-related disease are highly prevalent among persons with opioid use disorders (OUD). Unfortunately, traditional evidence-based smoking cessation interventions have yielded low rates of tobacco abstinence in this group. The majority of trials evaluating smoking cessation treatment interventions among persons with OUD have relied on short-term interventions that do not account for the unique challenges faced by these smokers, specifically, establishing initial abstinence, adhering to evidence-based cessation treatments, and maintaining abstinence once active treatments cease. Long-term smoking cessation medication treatment approaches have shown promise in promoting cessation and decreasing relapse among individuals without OUD, however the applicability of extended medication approaches to smokers with OUD may be limited by poor adherence to smoking cessation medications. Though adherence to cessation medication is strongly associated with cessation success, adherence is especially challenging for persons with OUD. Opioid treatment program-based directly observed therapy (DOT) interventions improve clinical outcomes in HIV and TB, and pilot data suggest that DOT varenicline is associated with increased smoking cessation medication adherence and may increase smoking cessation rates. In this 2 x 2 factorial, randomized, double-blind, placebo-controlled trial, the investigators will test two interventions: directly observed medication therapy, and long-term therapy with varenicline. The analytic strategy will evaluate the milestones in smoking cessation-achieving initial abstinence, preventing lapse and preventing relapse--necessary for long-term cessation, and evaluate theoretically-guided psychological and social factors and pharmacogenetic factors that influence these cessation processes. The investigators will recruit smokers with OUD from community-based, outpatient opioid treatment programs and test the following specific aims: (1) to test the efficacy of directly observed varenicline therapy compared to self-administered varenicline therapy on smoking cessation milestones, (2) to test the efficacy of long-term varenicline compared to short-term varenicline on smoking cessation milestones, and (3) to understand the mechanism of smoking cessation by examining the impact of theory-guided psychological and social factors and of pharmacogenetic factors on cessation milestones.

ELIGIBILITY:
Inclusion Criteria:

1) age ≥18 years old; 2) English or Spanish speaking (i.e., be able to participate in study interviews in English or Spanish); 3) current cigarette smoking (smoked at least 100 cigarettes/lifetime, smoking ≥ 5 cigarettes/day); 4) interest in quitting tobacco smoking; 5) receiving methadone or buprenorphine in the DoSA clinic one to six times weekly; 6) enrollment in a DoSA opioid treatment program ≥ 3 months; 7) stable methadone or buprenorphine dose for two weeks; 8) agreement to use contraception for the duration of the trial (among women with reproductive potential); 9) willingness to participate in all study components; and 10) ability to provide informed consent.

Exclusion Criteria:

1) serious or unstable disease, specifically: decompensated cirrhosis (INR≥ 1.7, albumin <2.7 g/dl or physical exam evidence of decompensated cirrhosis); severe cardiovascular disease (MI, PTCA, unstable angina, CABG, and/or serious arrhythmia in the previous 6 months); severe asthma or chronic obstructive pulmonary disease (requiring supplemental oxygen or hospitalization in past 6 months); HIV/AIDS (AIDS-defining illness or hospitalization in past 6 months); 2) creatinine clearance <30 mL/min; 3) history of seizure disorder; 4) women who are pregnant, breastfeeding, or contemplating pregnancy; 5) current suicidal ideation; 6) history of suicide attempt in the past year; 7) psychiatric hospitalization in the past year; 8) current DSM V criteria for major depressive episode, current bipolar disorder, or current psychotic disorder; 9) current DSM V criteria for alcohol use disorder; or 10) use of varenicline in the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Time-to-initial abstinence | Up to 24 weeks
  Time-to-initial abstinence, defined as a 24 hour period without smoking, will be assessed as Period of ≥ 24 hour self-reported abstinence during the intervention period, will be assessed. Group mean time-to-initial abstinence will be reported.
Time-to-lapse | Up to 24 weeks
  Time-to-lapse, defined as the initial occasion of cigarette smoking after abstinence, will be based on the first day during which subjects smoke, even a puff, after a period of initial abstinence. Group mean number of days to time-to-lapse will be reported.
Time to relapse | Up to 24 weeks
  Time-to-relapse, defined as the return to regular cigarette use, will be based on the time first day of seven consecutive days of self-reported smoking after a period of initial abstinence. Group mean number of days to time-to-relapse will be reported.

SECONDARY OUTCOMES:
Durability of 7-day point prevalence tobacco abstinence | week 28
  Durability of tobacco abstinence will be assessed using Carbon Monoxide (CO)-verified, 7-day point prevalence abstinence at week 28. Smoking abstinence in accordance with self-reported Timeline Follow Back Method (TLFB), which uses calendar prompts to assess self-reported daily patterns, and verified by expired carbon monoxide (CO) < 8 ppm, will be reported.
Durability of 7-day point prevalence tobacco abstinence | week 52
  Durability of tobacco abstinence will be assessed using Carbon Monoxide (CO)-verified, 7-day point prevalence abstinence at week 52. Smoking abstinence in accordance with self-reported Timeline Follow Back Method (TLFB), which uses calendar prompts to assess self-reported daily patterns, and verified by expired carbon monoxide (CO) < 8 ppm, will be reported.
Number of Cigarettes smoked per day | 24 weeks
  Group mean of self-reported number of cigarettes smoked per day will be obtained via self-reported TLFB and summarized per group.
Nicotine dependence | 24 weeks
  Nicotine dependence will be assessed using Fagerström Test of Nicotine Dependence (FTND). FTND is a 6-item instrument designed to provide an ordinal measure of nicotine dependence related to cigarette smoking. Specifically, the FTND evaluates the quantity of cigarette consumption, the compulsion to use, and dependence. Three Yes/No items are scored as either 0 (No) or 1 (Yes). Two multiple-choice items are either scored from 0-3 or 1-3, with higher scores signifying greater nicotine dependence. A final question, "Which cigarette would you hate to give up?" with 'First in the Morning' scored as 1 and 'Any other' scored as 0. The FTND yields an overall score of 0-10. An overall score of 1-2 = "Lowest Dependence", 3-4 = "Low to Moderate Dependence", 5-7 = "Moderate Dependence", and 8+ = "High Dependence"
Quality of life - Physical and Mental Health (SF-36) | 24 weeks
  Quality of Life will be assessed using the Medical Outcomes Study Short Form 12 (SF-12). The SF-12 is a 12-item general health questionnaire, derived from the Medical Outcomes Study 36 item Short Form Survey (SF-36), is designed to have similar performance as the SF-36, while taking less time to complete. The SF-12 asks a series of questions measuring eight health domains assessing both physical (PCS-12) and mental health (MCS-12). Two summary scores are generated: a mental component score (MCS-12), and a physical component score (PCS-12). Scores for both range from 0-100 with higher scores indicating better physical and mental health functioning, respectively. A score of 50 or less on the PCS-12 has been recommended as a cut-off to determine a physical condition, while a score of 42 or less on the MCS-12 may be indicative of 'clinical depression'. Group mean scores will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Shadi Nahvi, MD, MS, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Our final dataset will include: survey and laboratory data, including demographic, medical, tobacco, and other substance use-related information about all clinical trial subjects. The final dataset will be stripped of all personal identifiers.
Supporting Information: Study Protocol, Analytic Code
Time Frame: After data collection and cleaning is complete.
Access Criteria: We will share data with qualified investigators whose research protocols have been approved by their institutions' Institutional Review Boards. Data will be made available to potential users under a NIDA-approved data-sharing agreement that ensures that: (1) data is used only for research purposes and does not identify individual participants; (2) data is handled in a secure and confidential way; and (3) data is destroyed or returned after analyses are completed.